CLINICAL TRIAL: NCT01003808
Title: IMF-001 Phase 1 Study With Refractory Esophageal Tumor
Brief Title: Safety Study of a Recombinant Protein Vaccine to Treat Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoFrontier, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMF001J
Record Dates: First submitted 2009-10-16; First posted 2009-10-29 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMF-001 (Experimental): 100 or 200 mcg, subcutaneously every 2 weeks. Number of Injections: 6 times. (The treatment may be continued if it is beneficial to the subject).
  Interventions: Biological: IMF-001

INTERVENTIONS:
Biological: IMF-001 — 100 or 200 mcg, subcutaneously every 2 weeks. Number of Injections: 6 times. (The treatment may be continued if it is beneficial to the subject).
  Other Names: CHP-NY-ESO-1

SUMMARY:
The purpose of this study is to determine the biological recommended dose of IMF-001.

DETAILED DESCRIPTION:
The prognosis of esophageal cancer is improved with the improvement of surgery, chemotherapy and radiation therapy. However, there are no standard therapies established for recurrent esophageal cancer. NY-ESO-1 antigen is expressed in 33% of patients. NY-ESO-1 protein is applicable without limitation by HLA types, and injected as a complex with cholesteryl pullulan (CHP), forming nano-particles (IMF-001), it can activate both CD4+ and CD8+ T cells. In this phase 1 study, the safety and the biological recommended dose will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Radically unresectable stage III/IV esophageal tumors that have failed the standard treatment (including chemotherapy and radiotherapy), recurrent metastasis after radical surgery and not responding to the standard treatments, or recurrent metastasis after radiotherapy before/after radical surgery.
* Primary esophageal tumors confirmed by pathological diagnosis
* Tumor cells expressing NY-ESO-1 antigen (by tissue-immunostaining method or quantitative RT-PCR method)
* Performance status (PS) of 0, 1 or 2 (ECOG Scale)
* Life expectancy >/= 4 months
* No serious disorders with major organs (bone marrow, heart, lung, liver and kidney) and meets the following criteria:

  * WBC count >/= 2.0 x 10 9/L
  * Hemoglobin >/=8.0g/dL
  * Platelet count >/=75 x 10 9/L
  * Serum total bilirubin: </=1.5 x ULN (3 x ULN if with liver mets)
  * AST and ALT: </=2.5 x ULN (5x ULN if with liver mets)
  * Serum creatinine: </=1.5x ULN
* Agree to use birth control including condoms from the time of obtaining the consent to 6 months after the final administration of the study drug [except females after menopause (1 year or more after the last menstruation and females/males after an operation for sterilization)]
* Given written informed consent

Exclusion Criteria:

* HIV antibody positive
* Double cancer
* History of autoimmune disease
* History of severe anaphylaxis
* Active metastatic disease in the central nervous system (CNS) Within 4 weeks after treatment with an anti-tumor agent, systemically administered adrenocorticosteroids, immune suppressants or immune enhancers
* Pregnant or lactating
* Any other inadequacy for this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the maximum tolerated dose, dose-limiting toxicities, type/frequency/degree of adverse events and NY-ESO-1 antigen-specific immune response of IMF-001 alone in patients with esophageal cancer. | First 12 weeks (during the first 6 injections)

SECONDARY OUTCOMES:
To evaluate clinical activity (tumor response and time to progression). | Up to 2 years, or until progression of PS or no positive immune response from IMF-001.

CONTACTS AND LOCATIONS:
Overall Officials: Daiju Ichimaru, BSc, Study Director — ImmunoFrontier, Inc.
Locations (4):
- Japan (4):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Mie University Hospital, Tsu, Mie-ken
  - Kitano Hospital, Kitano Hospital, Osaka
  - Osaka University Hospital, Suita, Osaka

REFERENCES:
- [Background] Aoki M, Ueda S, Nishikawa H, Kitano S, Hirayama M, Ikeda H, Toyoda H, Tanaka K, Kanai M, Takabayashi A, Imai H, Shiraishi T, Sato E, Wada H, Nakayama E, Takei Y, Katayama N, Shiku H, Kageyama S. Antibody responses against NY-ESO-1 and HER2 antigens in patients vaccinated with combinations of cholesteryl pullulan (CHP)-NY-ESO-1 and CHP-HER2 with OK-432. Vaccine. 2009 Nov 16;27(49):6854-61. doi: 10.1016/j.vaccine.2009.09.018. Epub 2009 Sep 15. PMID 19761832
- [Background] Harada N, Hoshiai K, Takahashi Y, Sakaguchi Y, Kuno T, Hishida T, Shiku H. Preclinical safety pharmacology study of a novel protein-based cancer vaccine CHP-NY-ESO-1. Kobe J Med Sci. 2008 May 23;54(1):E23-34. PMID 18772606
- [Background] Tsuji K, Hamada T, Uenaka A, Wada H, Sato E, Isobe M, Asagoe K, Yamasaki O, Shiku H, Ritter G, Murphy R, Hoffman EW, Old LJ, Nakayama E, Iwatsuki K. Induction of immune response against NY-ESO-1 by CHP-NY-ESO-1 vaccination and immune regulation in a melanoma patient. Cancer Immunol Immunother. 2008 Oct;57(10):1429-37. doi: 10.1007/s00262-008-0478-5. Epub 2008 Mar 1. PMID 18311489
- [Background] Uenaka A, Wada H, Isobe M, Saika T, Tsuji K, Sato E, Sato S, Noguchi Y, Kawabata R, Yasuda T, Doki Y, Kumon H, Iwatsuki K, Shiku H, Monden M, Jungbluth AA, Ritter G, Murphy R, Hoffman E, Old LJ, Nakayama E. T cell immunomonitoring and tumor responses in patients immunized with a complex of cholesterol-bearing hydrophobized pullulan (CHP) and NY-ESO-1 protein. Cancer Immun. 2007 Apr 19;7:9. PMID 17441676
- [Background] Kawabata R, Wada H, Isobe M, Saika T, Sato S, Uenaka A, Miyata H, Yasuda T, Doki Y, Noguchi Y, Kumon H, Tsuji K, Iwatsuki K, Shiku H, Ritter G, Murphy R, Hoffman E, Old LJ, Monden M, Nakayama E. Antibody response against NY-ESO-1 in CHP-NY-ESO-1 vaccinated patients. Int J Cancer. 2007 May 15;120(10):2178-84. doi: 10.1002/ijc.22583. PMID 17278093
- [Background] Hasegawa K, Noguchi Y, Koizumi F, Uenaka A, Tanaka M, Shimono M, Nakamura H, Shiku H, Gnjatic S, Murphy R, Hiramatsu Y, Old LJ, Nakayama E. In vitro stimulation of CD8 and CD4 T cells by dendritic cells loaded with a complex of cholesterol-bearing hydrophobized pullulan and NY-ESO-1 protein: Identification of a new HLA-DR15-binding CD4 T-cell epitope. Clin Cancer Res. 2006 Mar 15;12(6):1921-7. doi: 10.1158/1078-0432.CCR-05-1900. PMID 16551878
- [Derived] Kageyama S, Wada H, Muro K, Niwa Y, Ueda S, Miyata H, Takiguchi S, Sugino SH, Miyahara Y, Ikeda H, Imai N, Sato E, Yamada T, Osako M, Ohnishi M, Harada N, Hishida T, Doki Y, Shiku H. Dose-dependent effects of NY-ESO-1 protein vaccine complexed with cholesteryl pullulan (CHP-NY-ESO-1) on immune responses and survival benefits of esophageal cancer patients. J Transl Med. 2013 Oct 5;11:246. doi: 10.1186/1479-5876-11-246. PMID 24093426